CLINICAL TRIAL: NCT03372135
Title: Postoperative Cognitive Deficit After Steep Trendelenburg Position and CO2 Pneumoperitoneum With Cerebral Oxygen: A Prospective Observational Pilot Study
Brief Title: Assessment of POCD After Steep Trendelenburg Position and CO2 Pneumoperitoneum With Cerebral Oxygen
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YYL
Record Dates: First submitted 2017-11-01; First posted 2017-12-13 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: POCD; RARC; Trendelenburg Position
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trendelenburg group: Patients in trendelenburg group take trendelenburg position and have CO2 pneumoperitoneum. Cerebral oxygen monitor will be needed. Take notes per hour for HR, MAP, CVP, SpO2, SrO2 and etCO2.Preoperative and postoperative ABG, S-100beta , CRP and cognitive dysfunction scales will be tested.
- Control group: Patients in control group take horizontal position. Cerebral oxygen monitor will be needed. Take notes per hour for HR, MAP, CVP, SpO2, SrO2 and etCO2.Preoperative and postoperative ABG, S-100beta , CRP and cognitive dysfunction scales will be tested

SUMMARY:
Postoperative cognitive decline (POCD) is a common and impactful outcome of surgical procedures in older adults. The pathophysiology and causative mechanisms for POCD are poorly understood. The robot-assisted radical cystectomy (RARC) is increasingly utilized. In patients undergoing RARC, Although prolonged Trendelenburg position and pneumoperitoneum can increase the cerebral blood flow, the excessive cerebral perfusion can lead to encephalemia, which reduce the oxygen uptake of brain tissue and cause insufficient oxygenation of brain tissue at the cellular level. POCD may take place due to cerebral hemodynamic changes. The goal of the current study is to investigate the combined effect of this position and CO2 pneumoperitoneum on POCD during RARC with the monitor of cerebral oxygen.

DETAILED DESCRIPTION:
Postoperative cognitive decline (POCD) is a short-term decline in cognitive function (especially in memory and executive functions) that may last from a few days to a few weeks after surgery. It is a common and impactful outcome of surgical procedures in older adults. The pathophysiology and causative mechanisms for POCD are poorly understood. It is supposed to be associated with numerous factors such as ages, trauma, inflammation, surgical stress, position, fluid, MBP, artificial pneumoperitoneum , PCO2, FiO2.

The robot-assisted radical cystectomy (RARC) is increasingly utilized. In patients undergoing RARC, Although prolonged Trendelenburg position and pneumoperitoneum can increase the cerebral blood flow, there were studies showed that the excessive cerebral perfusion can lead to encephalemia, which reduce the oxygen uptake of brain tissue and cause insufficient oxygenation of brain tissue at the cellular level. POCD may take place due to cerebral hemodynamic changes. Contemporary, intraoperative fluid restriction, a relatively long time of operation and surgical stress may also contribute to POCD.

The goal of the current study is to investigate the combined effect of this position and CO2 pneumoperitoneum on POCD during RARC with the monitor of cerebral oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Above age of 55
* Will undergo the robot-assisted radical cystectomy
* informed consent, volunteered to participate in this experiment, ASA I - III

Exclusion Criteria:

* Audio and visual impairment, illiteracy
* Existing severe central nervous system disease
* Patients with central nervous system disease or surgery , resulted in severe sequelae
* Alcohol dependence
* Take psychotropic medications
* Preoperative MMSE score was less than 24

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Chinese
Study Population: The study choose Chinese patients(ASA I - III
  ) above the age of 55, who will recently undergo the robot-assisted radical cystectomy. All those patients should be informed consent and be volunteered to participate in this experiment.
  Those audio and visual impairment, illiteracy,existing severe central nervous system disease, patients with central nervous system disease or surgery which resulted in severe sequelae, alcohol dependence, usage of psychotropic medications, reoperative MMSE score was less than 24 should be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of postoperative cognitive dysfunction | One week after surgery
  Using Z score method to analyse and comprehensively evaluate cognitive dysfunction scale which can help diagnosing the incidence of POCD.

SECONDARY OUTCOMES:
Probable risk factors of POCD | 1 year
  Diagnose and screen out patients with POCD and then analyse probable factors such as MAP, CVP, trendelenburg position etc as assesed by hierarchical regression analysis.
The effect of steep Trendelenburg position and CO2 Pneumoperitoneum on POCD | 1 year
  Comparison of morbidity is made between patients underwent RARC and those who have taken surgery in horizontal position.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Chen, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583
- [Background] Gainsburg DM. Anesthetic concerns for robotic-assisted laparoscopic radical prostatectomy. Minerva Anestesiol. 2012 May;78(5):596-604. Epub 2012 Mar 13. PMID 22415437
- [Background] Ding LL, Zhang H, Mi WD, Liu J, Jin CH, Yuan WX, Liu Y, Ni LY, Bo LL, Deng XM. [Anesthesia management of laparoscopic radical cystectomy and orthotopic bladder surgery with a robotic-assisted surgical system]. Beijing Da Xue Xue Bao Yi Xue Ban. 2013 Oct 18;45(5):819-22. Chinese. PMID 24136286
- [Derived] Li Y, Huang D, Su D, Chen J, Yang L. Postoperative cognitive dysfunction after robot-assisted radical cystectomy (RARC) with cerebral oxygen monitoring an observational prospective cohort pilot study. BMC Anesthesiol. 2019 Nov 6;19(1):202. doi: 10.1186/s12871-019-0877-5. PMID 31694553